CLINICAL TRIAL: NCT05244200
Title: The Impact of Insulin Staging in the Context of Pharmaceutical Care on Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Insulin Staging in the Context of Pharmaceutical Care on Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Kawa Ahmad Obeid, Head of the Department of Clinical Pharmacy., University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: College of Pharmacy/ UoS
Record Dates: First submitted 2022-01-07; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus.; Insulin Staging.; Pharmaceutical care.
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pharmaceutical Services

STUDY DESIGN:
Intervention Model Description: In these selective control trial, 100 patients with type 2 diabetes mellitus, those that they are on the end stage management protocol are going to be randomly allocated into two different groups, namely intervention and non-intervention groups. In the intervention group, a strict protocol developed by IDC for insulin prescription is going to be implement and patients will be assessed for the therapeutic outcomes along with the detection and resolution of drug therapy problems throughout the course of 6 months study. On the side, patients in the non-intervention group will be followed for the therapeutic outcomes and detection of DTPs without tempting to resolve them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Intervention Group (No Intervention): Patients in the non-intervention group will be followed for the therapeutic outcomes and detection of DTPs without tempting to resolve them
- Intervention Group (Experimental): A strict protocol developed by IDC for insulin prescription is going to be implement and patients will be assessed for the therapeutic outcomes along with the detection and resolution of drug therapy problems throughout the course
  Interventions: Other: Pharmaceutical care and insulin staging.

INTERVENTIONS:
Other: Pharmaceutical care and insulin staging. — Pharmaceutical care is a patient-centered practice in which the practitioner assumes responsibility for a patient's drug-related needs and is held accountable for this commitment. Due to the progressive nature of Type 2 Diabetes Mellitus, which requires timely optimization of treatment, leading in a majority of cases to insulin therapy, so that proper use of insulin is one of the critical tools for prevention of long-term complications. From the hundred patients in this study, half of the patients will be the control group without any intervention, and pharmaceutical care and insulin staging will be applied on the remaining. In this research two strategies will be applied including pharmaceutical care process and Insulin Staging approach on patients with T2DM, those who are on end stage treatment.
  Arms: Intervention Group

SUMMARY:
The number of people with diabetes rose from 108 million in 1980 to 422 million in 2014. Diabetes is a major cause of blindness, kidney failure, heart attacks, stroke and lower limb amputation. Current challenges in diabetes management include: (1) optimizing the use of currently available therapies to ensure adequate glycemic control and to reduce complications; (2) educating patients on diabetes self-management; (3) improving patient adherence to lifestyle and pharmacologic interventions; ; and (4) reducing barriers to the early use of insulin. In this research, the impact of pharmaceutical care and Insulin staging will be evaluated in patients with type 2 diabetes to overcome this challenges. The concept of "pharmaceutical care" was first introduced by Helper and Strand in 1990, pushing for the transformation of the Pharmacy profession from "product-focused" to "patient-centric". Pharmaceutical care is a patient-centered practice in which the practitioner assumes responsibility for a patient's drug-related needs and is held accountable for this commitment. Due to the progressive nature of the disease, which requires timely optimization of treatment, leading in a majority of cases to insulin therapy, so that proper use of insulin is one of the critical tools for prevention of long-term complications. From the hundred patients in this study, half of the patients will be the control group without any intervention, and pharmaceutical care and insulin staging will be applied on the remaining. In this research two strategies will be applied including pharmaceutical care process and Insulin Staging approach on patients with T2DM, those who are on end stage treatment.

DETAILED DESCRIPTION:
* In 2018, 34.2 million Americans, or 10.5% of the population, had diabetes.
* Of the 34.2 million adults with diabetes, 26.8 million were diagnosed, and 7.3 million were undiagnosed
* The percentage of Americans age 65 and older remains high, at 26.8%, or 14.3 million seniors (diagnosed and undiagnosed).
* Diabetes Mellitus (DM) is a group of metabolic disorders characterized by hyperglycemia and abnormalities in carbohydrate, fat, and protein metabolism.
* It results from defects in insulin secretion, insulin sensitivity, or both. Chronic microvascular, macrovascular, and neuropathic complications may ensue .
* One of the challenges facing the management of T2DM is the lack of an established guideline for Insulin administration in most of the communities.
* Considering the slogan of clinical pharmacy: safe, cost-effectiveness of medication, there are many Insulin products available and often doctors get confused on Choosing the right drug for the right patient.
* The hypothesis of this study is that clinical pharmacist Intervention through applying Pharmaceutical care and insulin staging has significant impact on quality of life and therapeutic outcomes of patients with Type II Diabetes With the end stage management protocol, while the null hypothesis states that there is no correlation between clinical pharmacist intervention with patient's quality of life and therapeutic outcomes.
* Study design: two-arm randomized, selective control trial.
* Interventions: Insulin Staging in the context of Pharmaceutical Care.
* Number of participants = 100.
* Number of groups = 2 groups each of 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* T2DM patients.
* Patients must be on insulin therapy
* Willing to participate in the study

Exclusion Criteria:

* T1DM
* T2DM patients whose not on insulin therapy
* Patients that have disabilities that interfere with compliances towards medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Mean change of glycated hemoglobin (HbA1c). | Up to 6 months.
  HbA1c refers to glycated hemoglobin (A1c) , which identifies average plasma glucose concentration (in %).
Measurement of Lipid profile (LDL, HDL, cholesterol and triglyceride) | Up to 6 months.
  Lipid profile refers to pattern of lipids in the blood (in mg/dL). A lipid profile usually includes the levels of total cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides, and the calculated low-density lipoprotein (LDL) 'cholesterol.
Measurement of Drug therapy problems (DTP). | Up to 6 months.
  Drug therapy problem (DTP) refers to any unwanted incident related to medication therapy that actually or potentially affects the desired goals of treatment.
Fasting plasma glucose (FPG) | Up to 6 months.
  FPG measures the levels of glucose in the plasma (in mg/dL).To assess the effect of insulin on the FPG level.

SECONDARY OUTCOMES:
Body Weight. | Up to 6 months.
  Body Weight: the amount that a person weighs (in kg), To find out whether the patient is obese or not.

CONTACTS AND LOCATIONS:
Overall Officials: Kawa Obeid, PhD, Principal Investigator — Clinical Pharmacy Department/ College of Pharmacy/University of Sulaimani/ Kurdistan Region-Iraq.
Locations (1):
- College of Pharmacy-University of Sulaimani, Sulaymaniyah, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whittlesea C, Hodson K. Clinical pharmacy and therapeutics. Elsevier 2019.
- [Background] Saseen JJ, Ripley TL, Bondi D, Burke JM, Cohen LJ, McBane S, McConnell KJ, Sackey B, Sanoski C, Simonyan A, Taylor J, Vande Griend JP. ACCP Clinical Pharmacist Competencies. Pharmacotherapy. 2017 May;37(5):630-636. doi: 10.1002/phar.1923. Epub 2017 May 2. PMID 28464300
- [Background] Cipolle RJ, Strand LM, Morley PC. Pharmaceutical care practice: the clinician's guide. 2nd ed. New York: McGraw-Hill, Medical Pub. Division; 2004. 394 p.
- [Background] Chumney EC, Robinson LC. The effects of pharmacist interventions on patients with polypharmacy. Pharm Pract (Granada). 2006 Jul;4(3):103-9. PMID 25247007
- [Background] Mansour A, Al Douri F. Diabetes in Iraq: Facing the Epidemic. A systematic Review. Wulfenia. 2015;22(3):258.